CLINICAL TRIAL: NCT06863090
Title: A Single-centre Feasibility Study Investigating the Use of in Vivo Dosimetry in Patients Receiving High Dose Rate (HDR) Brachytherapy for Gynaecological and Prostate Cancers
Brief Title: In Vivo Dosimetry for Brachytherapy Study
Status: Recruiting | Type: Observational
Sponsor: East and North Hertfordshire NHS Trust (Other Government)
Collaborators: TRUEinvivo Limited (Unknown)
Responsible Party: Sponsor
Other Study IDs: RD2024-15
Record Dates: First submitted 2025-03-03; First posted 2025-03-07 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Prostate Cancer; Gynaecological Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Prostate cancer patients: histologically proven primary or recurrent prostate cancer
- Gynaecological cancer patient: locally advanced gynaecological malignancy in the primary and recurrent setting

SUMMARY:
The main study aim is the investigate the clinical use of in vivo dosimeters (small measurement devices) for brachytherapy (internal radiotherapy).

DETAILED DESCRIPTION:
A dosimeter is a small device that is able to record the dose of radiation received. It can provide an independent check that the dose of radiation delivered matches the dose calculated for patients receiving radiotherapy as part of their cancer treatment.

The purpose of this study is to investigate the clinical use of in vivo dosimeters for brachytherapy. Two types of dosimeters will be used; micro metal oxide field effect transistors (microMOSFETs) and Thermoluminescent detectors (TLDs). These will be placed into the rectum (back passage), urethra (the tube through which urine leave the body from the bladder) and within or near (typically within a few centimetres) to the cancer itself. These devices will record the dose of radiation received at the time of brachytherapy at each of these sites and we will compare that measurement with the expected measurement based on the calculations we made in planning the patient's treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and above
* Patients receiving HDR brachytherapy using iridium-192 (192Ir) radioactive source either as a monotherapy or in combination with external beam radiotherapy for:

  1. histologically/radiologically proven primary or locally recurrent prostate cancer
  2. locally advanced gynaecological malignancy in the primary and recurrent setting

     * primary cervix carcinoma (squamous, adenocarcinoma, adenosquamous) FIGO IB2-IVA
     * primary vulval FIGO I-IVA
     * primary vaginal FIGO I-IVA
     * primary endometrial cancer FIGO Stage I-IVA (not suitable for surgery)
     * endometrial cancer receiving adjuvant vaginal vault brachytherapy
     * recurrent cervix, vulval, vaginal or endometrial cancer suitable for brachytherapy as discussed in a regional gynae-oncology multidisciplinary meeting.
* World Health Organisation (WHO) or Eastern Cooperative Oncology Group (ECOG) performance status 0-2

Exclusion Criteria:

* Previous brachytherapy exposure to the treatment site
* Patients unable to give informed consent
* Patients unable to have a regional or general anaesthetic
* Patients with the following medical conditions: coagulopathies, history of another primary malignancy, known allergy or sensitivity to study materials; previous or current fistulae
* Not able to understand the implications of participating in the study in English
* Patients with recent (within the last 6 months) or currently participating in interventional research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving high dose rate (HDR) brachytherapy for gynaecological and prostate cancers
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-03-03 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
To assess the feasibility of in vivo dosimetry in HDR brachytherapy and compare the calculated dose against measured dose | 12 months
  Measured by comparing the calculated (treatment planning system (TPS)) dose against the measured dose (using micro silica thermo-luminescent dosimeters (TLDs) and micro metal oxide field effect transistors (MOSFETS)). The measured dose will be compared to the calculated dose by the TPS at the bladder neck, anterior rectal wall, recto-vaginal point (gynaecological cases) and within the clinical target volume (CTV) for each fraction as well for the whole treatment.

SECONDARY OUTCOMES:
Review of investigative and corrective action | 12 months
  Measured by defined action thresholds during high-dose rate (HDR) brachytherapy

CONTACTS AND LOCATIONS:
Overall Officials: Peter Hoskin, Principal Investigator — East and North Hertfordshire NHS Trust
Locations (1):
- Mount Vernon Cancer Centre, Northwood, Middlesex, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
The research results will be published in international journals and presented at scientific meetings.